CLINICAL TRIAL: NCT04363567
Title: Endothelial Glycocalyx Evaluated on Release of the Endothelial Glycocalyx Proteins and Salt Blood Test in Patients With Chronic Kidney Disease
Brief Title: Endothelial Glycocalyx in Patients With Chronic Kidney Disease
Acronym: EGNI
Status: Completed | Type: Observational
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Jesper Norgaard Bech, Chief Physician and PhD, Regional Hospital Holstebro
Other Study IDs: RLS-3-2016
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Healthy; Chronic Kidney Diseases
Keywords: Salt blood test; endothelial glycocalyx; chronic kidney disease; syndecan-1; heparan sulfate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- CKD 1: Patients with Chronic kidney disease stage 1: Normal kidney function but urine findings or structural abnormalities or genetic trait point to kidney disease. eGFR :90+.
  20 patients, maximun 4 patients with diabetes.
- CKD 2: Patients with Chronic kidney disease stage 2: Mildly reduced kidney function, and other findings (as for stage 1) point to kidney disease. eGFR: 60-89.
  20 patients, maximun 4 patients with diabetes.
- CKD 3: Patients with Chronic kidney disease stage 3: Moderately reduced kidney function. eGFR: 30-59.
  20 patients, maximun 4 patients with diabetes.
- CKD 4: Patients with Chronic kidney disease stage 4: Severely reduced kidney function. eGFR: 15-29.
  20 patients, maximun 4 patients with diabetes.
- CKD 5: Patients with Chronic kidney disease stage 5: Very severe kidney function. eGFR: <15.
  20 patients, maximun 4 patients with diabetes.
- Dialysis: Patients with end stage renal disease in dialysis. 20 patients, maximun 4 patients with diabetes.
- Healthy: 20 healthy people. Control group

SUMMARY:
The luminal side of the entire vasculature is covered with a gel-like polymer called endothelial glycocalyx (EG). EG is important for the transport of molecules in and out of the blood cells and for endothelial function. EG protects the blood vessel wall, is likely to contribute to maintenance of normal blood pressure and the prevention of blood clot formation. Overall it is likely to avoid development of cardiovascular disease.

A newly developed blood test, salt-blood test, can measure erythrocyte salt sensitivity and gives information about the condition of EG. EG can also be measured by release of endothelial glycocalyx proteins.

Previous studies indicate that this EG is impaired by a number of chronic diseases, including chronic kidney disease. This study investigates the quality of glycocalyx in patients with chronic kidney disease, and compares with the layer in healthy.

DETAILED DESCRIPTION:
The purpose of this study is to gain knowledge about how pronounced the EG are affected in varying degrees of chronic kidney disease compared with healthy controls assessed by

1. salt-blood test
2. release of endothelial glycocalyx proteins.

and to see how this correlates to

1. blood pressure (peripheral and central)
2. pulse wave velocity
3. albuminuria
4. coagulation system
5. vasoactive hormones (PRC, p-Ang-II, p-Aldo, p-ANP, p-BNP, p-AVP)

ELIGIBILITY:
Inclusion Criteria patients with chronic kidney disease:

CKD I-V Age> 18 years 4 diabetics in each CKD-class Dialysis patients must have received dialysis for at least 3 months. Signed consent

Exclusion Criteria, patients with chronic kidney disease:

Nephrotic syndrome (U-alb> 3.5 g / d, p-alb <30 g / l, and peripheral edema) Alcohol abuse Drug abuse Pregnancy and lactation Hbg <6.2 mmol / l

Inclusion criteria, healthy people:

Both gender Signed consent

Exclusion criteria, healthy people:

Arterial hypertension heart, lung, liver, kidney, endocrine og cerebral diseases alcohol, drug or medical abuse smoking pregnancy or breastfeeding blood-donation within a month clinically significant abnormalities in ECG, blood samples or urine samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidneys disease in different stages and healthy volunters as control group.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Erythrocyte Salt Sensitivity | 1 minute
  Blood sample

SECONDARY OUTCOMES:
Syndecan-1 | 1 minute
  blood sample
Heparan Sulfate | 1 minute
  blood sample
blood pressure central and peripheral | 1 minute
  Mobil-O-Graph
Vasoactive hormones (PRC, Ang-II, Aldo, ANP, BNP, AVP) | 1 minute
  blood samples
pulse wave velocity | 1 minute
  Mobil-O-Graph
Albuminuria | 1 minute
  urine sample
coagulation | 1 minute
  blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Lu Sønderbæk, MD, Principal Investigator — Department of medical research and medicine

IPD SHARING:
Plan to Share IPD: No